CLINICAL TRIAL: NCT01384344
Title: Ecological Assessment of Apathy in Alzheimer's Disease and in Control Subjects: Interest on Video Recognition and Actigraphy
Brief Title: Ecological Assessment of Apathy in Alzheimer's Disease and in Control Subjects: Video Recognition and Actigraphy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 11-PP-03
Record Dates: First submitted 2011-05-27; First posted 2011-06-29 (Estimated); Last update posted 2012-12-18 (Estimated); Status verified 2011-05

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Watchful Waiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- witness (Active Comparator): no mnesic complaint
  Interventions: Other: observational
- Alzheimer disease with apathy (Experimental): Alzheimer's disease according to criteria of NINCDS-ADRDA with apathy
  Interventions: Other: observational
- Alzheimer's disease without apathy (Experimental): Alzheimer's disease according to criteria of NINCDS-ADRDA without apathy
  Interventions: Other: observational

INTERVENTIONS:
Other: observational — Observation during a physical exercise

SUMMARY:
Cognitive and memory disorders are characterized of Alzheimer disease. In addition, psychologic and behavioural symptoms, called speak neuropsychiatric symptoms, are frequents and play an important role in prognostic and intervention. These symptoms are noticed before the diagnostic of dementia, their prevalence and their intensity increase with the evolution of disease. Apathy, which is characterized by a decrease of motivation, is the most frequent of this behaviour disrupt. Clinically, a decrease, or a totally, lack of interest, initiative and blunting emotional are noticed. Fundamentally, apathy is considered as a decrease of cognition and behaviour to "go in goal". Assessment of psychological and behavioural symptoms is realised principally with neuropsychiatric scales. These contribute to obtain particular informations about health of patient allowing by patient and caregiver discussions and impressions of clinician. These scales are simples but loss of subjectivity. An alternative of this method is the use of gerontechnology as actigraphy (system out-patient which records locomotive activity with the help of piezo-electrical sensor fixed on a bracelet) and video recording which is associated to an informatic treatment of signal in order event recognition.

The aim of study is to realise an objective assessment of activities "go in goal" during experimental sequence which has well-characterized acts, using at the same time an actigraphic record of activity "motive" (system of assessment indirect of apathy fit) and a video records which uses an informatic event recognition system. The assessment will realise with participants controls (n=30) and Alzheimer disease patients with (n=20) or without (n=20) apathy, during well-characterized records. The final aim is to obtain a particular assessment of some disorders behaviours, as apathy, which is principally characterize by a decrease of behaviours "to go in goal".

ELIGIBILITY:
Inclusion Criteria for no mnesic patient:

* man or female, more 65 years ;
* no caregiver ;
* no motor handicap ;
* no global cognitive impairment with > 26 MMSE, neither argument in favour of following diagnosis : Alzheimer's disease, major depressive episode ;
* no apathy ;
* participant with french national health ;
* signature of informed consent.

Inclusion Criteria for Alzheimer's patient:

* man or female, more 65 years ;
* no motor handicap ;
* with diagnosis of Alzheimer's disease according to criteria of NINCDS-ADRDA ;
* apathy score > 3 in Neuropsychiatric Inventory ;
* with a MMSE score lower than 26/30 ;
* with cholinesterase inhibitor medication, standard and stable dose since 3 month ;
* no global cognitive impairment with > 26 MMSE, neither argument in favour of following diagnosis : Alzheimer's disease, major depressive episode ;
* no apathy ;
* participant with french national health ;
* signature of informed consent.

Exclusion Criteria:

* Impossibility of realization of the experimental protocol because of a driving handicap.
* Port(Bearing) of a pacemaker
* Under guardianship Patient or guardianship

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 82 (Actual)
Dates: Start 2011-06; Primary Completion 2011-12 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
stride and speed walking | one time point - at the only visit of protocol (day 1)

SECONDARY OUTCOMES:
For comparison between Alzheimer disease patients with (n=20) or without apathy, we use again stride and speed walking | one time point - at the only visit of protocol (day 1)
For reproducibility, we use stride and speed walking | one time point - at the only visit of protocol (day 1)
Reliability is the sum of posture's concordance | one time point - at the only visit of protocol (day 1)
Relation between LF/HF variations and activity index | one time point - at the only visit of protocol (day 1)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe ROBERT, PU-PH, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- Hôpital de Cimiez, Nice, France